CLINICAL TRIAL: NCT06227897
Title: A Single-Arm, Open-Lable Study of Adjuvant Aumolertinib for Completely Resected Stage IB-IIIA Non-Small-Cell Lung Cancer With EGFR Exon 19 Deletion or L858R Mutations.
Brief Title: Aumolertinib in EGFR-Mutant Resected Stage IB-IIIA NSCLC (AERESA).
Acronym: AERESA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO10109
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
Keywords: Lung cancer, EGFR, adjuvant
MeSH Terms: conditions — Lung Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aumolertinib (Experimental): Aumolertinib 110 mg once daily (110 mg per day) orally for 36 months.
  Interventions: Drug: Aumolertinib

INTERVENTIONS:
Drug: Aumolertinib — Aumolertinib 110 mg per day orally for 3 years.
  Other Names: almonertinib; HS-10296

SUMMARY:
Aumolertinib (almonertinib; HS-10296) is a novel third-generation EGFR-TKI showing activity against EGFR-sensitizing mutations and EGFR T790M mutation. The third-generation EGFR-TKI osimertinib has been approved in the adjuvant setting. This study is to studying 3-year aumolertinib as adjuvant therapy to see how well it works in treating patients with resected stage IB-IIIA NSCLC harboring sensitizing EGFR mutations.

DETAILED DESCRIPTION:
Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) show great efficacy in patients with advanced non-small cell lung cancer (NSCLC) with EGFR mutations. Aumolertinib (almonertinib; HS-10296) is a novel third-generation EGFR-TKI. Aumolertinib showed activity against EGFR-sensitizing mutations and EGFR T790M mutation. In the phase III AENEAS trial, aumolertinib had improved efficacy to gefitinib with similar safety. In the phase II APOLLO trial, aumolertinib is effective and well-tolerated for patients with advanced NSCLC having an EGFR T790M mutation after disease progression on first- and second-generation EGFR TKI therapy. The third-generation EGFR-TKI osimertinib has been approved in the adjuvant setting. This study is to studying 3-year aumolertinib as adjuvant therapy to see how well it works in treating patients with resected stage IB-IIIA NSCLC harboring sensitizing EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

* Target population is high risk NSCLC with resection option for potential cure, as assessed by a faculty surgeon at SYSUCC. This may include clinical stage IB (≥4cm), II and IIIA. Subjects with N3 nodal involvement are not included.
* Subjects should have a detected sensitizing EGFR.
* Written informed consent provided.
* Male and female, aged 18-75 years.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Blood and specimens before and after treatment must be provided
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy ≥12 weeks.
* EGFR activating mutation in exon 19 or 21.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Known severe hypersensitivity to aumolertinib or any of the excipients of this product.
* Had had previous chemotherapy, radiotherapy, or agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Evidence of clinically active interstitial lung disease.
* Eye inflammation not fully controlled or conditions predisposing the subject to this.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* History of another malignancy in the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Patient who has active serious infection (e.g. pyrexia of or 38.0℃ over)
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Women who are pregnant or nursing.
* Ingredients mixed with small cell lung cancer patients.
* History of neurologic or psychiatric disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation.
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
3-year Disease Free Survival | 3 years after the last patient is randomized
  3-year DFS was defined as the proportion of patients who were disease free at 3 years.

SECONDARY OUTCOMES:
Disease Free Survival | 3 years
  Disease-free survival was assessed from randomization to disease recurrence or death as a result of any cause.
Adverse Events | 2 years after the last patient is randomized
  Adverse Events were monitored according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.
Number of participants with perioperative complications | 2 years
  Number of participants with perioperative complications
3-year Overall Survival | 3 years after the last patient is randomized
  3-year OS was defined as the proportion of patients who were alive at 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF